CLINICAL TRIAL: NCT05467826
Title: Efficacy and Safety of Sofosbuvir/Velpatasvir Plus Ribavirin for 12 Weeks or Sofosbuvir/Velpatasvir/Voxilaprevir for 12 Weeks in DAA Treatment Naïve HCV Subjects With GT3b, Compensated Cirrhosis in China
Brief Title: Efficacy and Safety of SOF/VEL + RBV and SOF/VEL/VOX for 12 Weeks in HCV Subjects With GT3b and Compensated Cirrhosis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Huiying Rao, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PKU-HCV-3B
Record Dates: First submitted 2022-07-18; First posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Hepatitis C; Cirrhosis
MeSH Terms: conditions — Hepatitis C; Fibrosis | interventions — Sofosbuvir; velpatasvir; Ribavirin; sofosbuvir-velpatasvir drug combination; sofosbuvir velpatasvir voxilaprevir drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Sofosbuvir 400mg/velpatasvir 100mg + ribavirin 1000mg/1200mg for 12 weeks
  Interventions: Drug: Sofosbuvir/Velpatasvir + Ribavirin
- Arm 2 (Experimental): Sofosbuvir 400mg/velpatasvir 100mg/voxilaprevir 100mg for 12 weeks
  Interventions: Drug: Sofosbuvir/Velpatasvir/Voxilaprevir

INTERVENTIONS:
Drug: Sofosbuvir/Velpatasvir + Ribavirin — Sofosbuvir 400mg/velpatasvir 100mg + ribavirin 1000mg/1200mg for 12 weeks
  Other Names: Epclusa
  Arms: Arm 1
Drug: Sofosbuvir/Velpatasvir/Voxilaprevir — Sofosbuvir 400mg/velpatasvir 100mg/voxilaprevir 100mg for 12 weeks
  Other Names: Vosevi
  Arms: Arm 2

SUMMARY:
Direct-acting antiviral agents (DAAs) targeting HCV have revolutionized the treatment of HCV. The efficacy of DAA-based therapy can depend on patient-related factors such as treatment experience, cirrhosis, but also on viral genotype. The high prevalence of genotype 3, which is considered difficult to cure, remains a challenge because many oral DAAs are less effective for this genotype, particularly subtype 3b than for others. Current guidance generally recommends sofosbuvir (SOF)/velpatasvir (VEL) ± ribavirin (RBV), glecaprevir/pibrentasvir and SOF/VEL/voxilaprevir (VOX) as first-line therapy for genotype 3, and an interferon-based regimen - SOF plus pegylated interferon and ribavirin is still recommended as an alternative treatment option. These recommendations are based on clinical data generated in regions where genotype 3a predominates. Our recent study indicated that sofosbuvir plus ribavirin for 24 weeks in subjects with HCV genotype 3 infection resulted in high rates of SVR. However, the SVR12 rate among subjects with genotype 3b was lower than that observed in subjects with genotype 3a infection, particularly among treatment-experienced subjects with cirrhosis.

Our study aimed to investigate the efficacy and safety of SOF/VEL plus RBV for 12 weeks or SOF/VEL/VOX for 12 weeks in DAAs treatment naïve HCV subjects with GT3b, compensated cirrhosis in China.

DETAILED DESCRIPTION:
Chronic hepatitis C virus (HCV) infection, which may lead to cirrhosis and hepatocellular carcinoma, is a major cause of chronic liver disease worldwide. Genotype 3 is the second most common genotype globally, accounting for approximately 18% of all adult HCV infections. Subjects with HCV genotype 3 infection, particularly genotype 3b, have a greater risk of developing hepatic steatosis, more rapid progression of hepatic fibrosis and cirrhosis, and hepatocellular carcinoma. Although there is only a small percentage of HCV subjects with genotype 3 in East Asia (5.4%) and China (8.7%), genotype 3b represents more than 50% of genotype 3 subjects in China,compared to most other regions of the world where genotype 3a predominates. In certain provinces of China, such as Yunnan Guizhou, and Chongqing, genotype 3b is the predominant HCV subtype among genotype 3 subjects.

Direct-acting antiviral agents (DAAs) targeting HCV have revolutionized the treatment of HCV. The efficacy of DAA-based therapy can depend on patient-related factors such as treatment experience, cirrhosis, but also on viral genotype. The high prevalence of genotype 3, which is considered difficult to cure, remains a challenge because many oral DAAs are less effective for this genotype, particularly subtype 3b than for others. Current guidance generally recommends sofosbuvir (SOF)/velpatasvir (VEL) ± ribavirin (RBV), glecaprevir/pibrentasvir and SOF/VEL/voxilaprevir (VOX) as first-line therapy for genotype 3, and an interferon-based regimen - SOF plus pegylated interferon and ribavirin is still recommended as an alternative treatment option. These recommendations are based on clinical data generated in regions where genotype 3a predominates. Our recent study indicated that sofosbuvir plus ribavirin for 24 weeks in subjects with HCV genotype 3 infection resulted in high rates of SVR. However, the SVR12 rate among subjects with genotype 3b was lower than that observed in subjects with genotype 3a infection, particularly among treatment-experienced subjects with cirrhosis.

Our study aimed to investigate the efficacy and safety of SOF/VEL plus RBV for 12 weeks or SOF/VEL/VOX for 12 weeks in DAAs treatment naïve HCV subjects with GT3b, compensated cirrhosis in China.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent
2. Male or female, age ≥18 years
3. Body mass index (BMI) between 18.0-35.0kg/m2 and bodyweight ≥ 40 kg
4. Chronic HCV infection (≥ 6 months) documented by prior medical history or liver biopsy
5. Anti-HCV positive at screening
6. HCV RNA 104 IU/mL at screening by the Central Laboratory
7. HCV genotype 3b assessed at screening by the Central Laboratory
8. DAA treatment naïve defined as having never been exposed to approved or experimental HCV-specific direct-acting antiviral agents. Pegylated interferon/interferon based prior treatment is allowed.
9. Cirrhosis Determination: cirrhosis is defined as any one of the following:

   1. Liver biopsy showing cirrhosis (e.g., Metavir score = 4 or Ishak score ≥5) in 24 months before screening, or
   2. Fibroscan® with a result of >12.5 kPa in 6 months before screening
10. The lab test at screening should meet all the criterion below: a) ALT ≤ 10 the upper limit of normal (ULN); b) AST ≤ 10 ULN; c) Total bilirubin ≤ 2 ULN; d) Platelets ≥ 60,000/L; e) Neutrophile ≥ 1,500/L; f) HbA1c ≤ 8.5%; g) Creatinine clearance (CLcr) ≥ 60 mL /min as calculated by the Cockcroft-Gault equation; h) Hemoglobin ≥ 11 g/dL for female subjects; ≥ 12 g/dL for male subjects; i) Albumin ≥ 3 g/dL; j) INR ≤ 1.7 x ULN; k) AFP <100ng/mL；if 20ng/mL≤AFP≤100ng/mL，HCC should be exclude by liver ultrasound
11. Females of childbearing potential must have a negative serum pregnancy test at screening
12. Male subjects and female subjects of childbearing potential who engage in heterosexual intercourse must agree to use protocol specified method(s) of contraception
13. Male subjects must agree to avoid donating sperm in 6 months after the last dose of drug
14. Subject must be of generally good health, with the exception of chronic HCV infection, as determined by the Investigator
15. Subject must be able to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments

Exclusion Criteria:

1. Decompensated cirrhosis, including but not limited to: prior or current ascites, variceal hemorrhage and/or hepatic encephalopathy; prior or current Child-Pugh B or C
2. HBsAg posititve at screening
3. Anti-HIV positive at screening
4. Alcohol abuse
5. Contraindication of ribavirin, including but not limited to hemoglobinapathy
6. Pregnant or nursing female or male with pregnant female partner
7. Use of any prohibited concomitant medications as described in Section before screening
8. Known hypersensitivity to SOF, VEL, RBV or formulation excipients
9. Subjects who has any of the following history: a) Chronic liver disease of a non-HCV etiology (e.g., hemochromatosis, Wilson's disease, alfa-1 antitrypsin deficiency, cholangitis); b) Solid organ transplantation; c) Significant pulmonary disease, significant cardiac disease or porphyria; d) Pancreatitis; e) Autoimmune diseases (e.g., systemic lupus erythematosus, sarcoidosis, psoriasis); f) Psychiatric hospitalization, suicide attempt, and/or a period of disability as a result of their psychiatric illness within the last 5 years; g) Malignancy within the 5 years prior to screening, with the exception of specific cancers that have been cured by surgical resection (basal cell skin cancer, etc). Subjects under evaluation for possible malignancy are not eligible; h) Significant drug allergy (such as anaphylaxis or hepatotoxicity).
10. Assessed as ineligible by investigators

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-09-01 (Estimated); Primary Completion 2023-11-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with SVR12 | 12 weeks post treatment.
  To evaluate the efficacy of treatment with SOF/VEL plus RBV for 12 weeks or SOF/VEL/VOX for 12 weeks in DAA treatment naïve HCV participants with GT3b, participants initiated on treatment will be assessed for viral load response at 12 weeks post treatment (SVR12). We use the proportion of participants with SVR12 as primary outcome measure.

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | Treatment start date through treatment completion (up to 24 weeks).
  Number of Participants With treatment-related adverse events as assessed by CTCAE v4.0- SOF/VEL plus RBV vs. SOF/VEL/VOX.

CONTACTS AND LOCATIONS:
Overall Officials: Huiying Rao, Dr., Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Huang R, Ji F, Jiang Y, Li S, Su M, Zhong Y, Zu H, Ding Y, Kong X, Shang J, Wei L, Rao H. Sofosbuvir/Velpatasvir/Voxilaprevir Versus Sofosbuvir/Velpatasvir Plus Ribavirin in Patients With Hepatitis C Virus Genotype 3b and Compensated Cirrhosis: A Multicentre Randomized Controlled Trial. J Med Virol. 2025 Nov;97(11):e70709. doi: 10.1002/jmv.70709. PMID 41255102